CLINICAL TRIAL: NCT05695170
Title: Couple-Based Lifestyle Intervention to Prevent Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Baucom, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 143079; K23DK115820 (NIH); 3K23DK115820-05S1 (NIH)
Record Dates: First submitted 2022-12-28; First posted 2023-01-23 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: PreDiabetes; Prediabetic State; Overweight and Obesity
Keywords: Lifestyle Intervention; Prevention; Social Support; Couple Relationships
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Nurses who assess health markers and behaviors pre programs will be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual intervention condition (Active Comparator): "PreventT2" individual lifestyle intervention curriculum (2021 revised National DPP curriculum, freely available from the CDC)
  Interventions: Behavioral: PreventT2 (Individual intervention)
- Couple-based intervention condition (Experimental): "PreventT2 Together" (couple-based adaptation of PreventT2; approved by the CDC in November 2022 as an Alternate Curriculum for use in the National DPP)
  Interventions: Behavioral: PreventT2 Together (Couple-based intervention)

INTERVENTIONS:
Behavioral: PreventT2 (Individual intervention) — PreventT2 will be delivered by a team of trained CDC Lifestyle Coaches to adults at high risk for diabetes. The 2021 version of the curriculum that will be used is freely available from the CDC. The intervention will be delivered in the context of the University of Utah National Diabetes Prevention Program (DPP), which has "full" recognition from the CDC based on outcome data over the course of a number of years.
  Arms: Individual intervention condition
Behavioral: PreventT2 Together (Couple-based intervention) — PreventT2 Together will be delivered by a team of trained CDC Lifestyle Coaches to adults at high risk for diabetes and their partners. The curriculum was developed with the input of a community advisory board and was approved by the CDC for use in the National DPP (i.e., meets CDC Diabetes Prevention Recognition Program Standards, including 22+ classes delivered over the course of 12 months and targeting lifestyle changes to prevention type 2 diabetes). In contrast to PreventT2, the intervention includes content specific to couples with prompts encouraging partners to consider and discuss how they can best support one another, information about lifestyle intervention in a relationship context, and examples demonstrating how couples collaborated to make healthy lifestyle changes.
  Arms: Couple-based intervention condition

SUMMARY:
The goal of this randomized pilot clinical trial is to describe the feasibility of a couple-based lifestyle intervention and the study protocol in preparation for a future definitive randomized clinical trial. Participants include individuals at risk for type 2 diabetes and their romantic partners.

The main objectives are:

1. To describe the feasibility of the couple-based intervention.
2. To describe the feasibility of the study protocol for use in a definitive trial.

Participating couples will be randomized to one of two year-long lifestyle intervention conditions: an individual curriculum or a couple-based curriculum.

Participants will complete assessments before and after the year-long intervention, as well as monthly during the intervention. Data will be collected on: feasibility, background, health behaviors, physical and mental health, and relationship functioning.

DETAILED DESCRIPTION:
The goal of this randomized pilot clinical trial is to describe the feasibility of a couple-based lifestyle intervention and the study protocol in preparation for a future definitive randomized clinical trial. Participants include individuals at risk for type 2 diabetes and their romantic partners.

Prior to all study procedures, eligible participants will be required to complete an informed consent process and electronically sign a consent document. 12 eligible couples will be randomly assigned to either an individual lifestyle intervention (PreventT2) or a couple-based adaptation designed with input from a community advisory board (PreventT2 Together) (1:1). Both curricula have CDC approval for use in the National DPP and are delivered to small groups of participants over the course of 12 months.

Across conditions, participants will complete assessments before and after the year-long intervention, as well as monthly during the intervention. Data will be collected on: feasibility, background, health behaviors, physical and mental health, and relationship functioning.

ELIGIBILITY:
Both the "target individual" (i.e., individual at high risk for type 2 diabetes) and "supporting partner" (i.e., partner of target individual) must meet eligibility criteria in order for a couple to enroll in the study.

* Eligibility criteria for "target individuals":

  1. Eligible for National DPP.

     A. DPP Inclusion Criteria:

  1) BMI of ≥ 25 kg/m2 (≥ 23kg/m2 if Asian) AND 2) High risk for type 2 diabetes, based on 1+ of the following three:
  1. CDC/American Diabetes Association Prediabetes Risk Test score ≥ 5
  2. Blood test results indicative of prediabetes in the past year (i.e., fasting blood glucose 100-125 mg/dl; blood glucose of 140-199 mg/dl 2 hours after a 75 g glucose load; OR 6.4% ≥ HbA1c ≥ 5.7%)
  3. Previous diagnosis of gestational diabetes (among women)

     B. DPP Exclusion Criteria:
     1. Diagnosis of type 1 diabetes or type 2 diabetes
     2. Currently pregnant

     AND

     2. Eligible for Study (Additional Criteria).

     A. Study Inclusion Criteria:
     1. Living together for 1+ year
     2. Report being in a romantic relationship
     3. Conversational fluency in English
     4. Age 18 or older
     5. Interested in participating

     B. Study Exclusion Criteria
     1. Diagnosis of another chronic disease (unless stable or with no major events/changes for 3+ months);
     2. Current medication for prediabetes or obesity;
     3. Current participation in lifestyle intervention for prediabetes or obesity;
     4. Past participation in the National DPP;
     5. Not comfortable participating in intervention together with partner.
* Eligibility criteria for "supporting partners":

A. Study Inclusion Criteria:

1. Partner meets "target individual" eligibility criteria (per above)
2. Living together for 1+ year
3. Report being in a romantic relationship
4. Conversational fluency in English
5. Age 18 or older
6. Interested in participating

B. Study Exclusion Criterion

1) Not comfortable participating in intervention together with partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Couple-based intervention feasibility | 1.5 years
  Participants will complete the Theoretical Framework of Acceptability-Based Questionnaire and two open-ended survey items developed by the research team monthly during the intervention and at post-intervention. Participants will also complete a post-intervention qualitative joint couple interview that utilizes a semi-structured couple interview guide. Lifestyle Coaches will also report on attendance, completion of weekly activity logs, and completion of make-up sessions.
  The team of Lifestyle Coaches delivering PreventT2 Together will also complete open-ended items developed by the research team following each class. Lifestyle Coaches will also complete a measure of barriers to participation and lifestyle change they observed among the participants, as well as several measures based on implementation outcomes (i.e., Acceptability of Intervention Measure, Intervention Appropriateness Measure, Feasibility of Intervention Measure).
Study protocol feasibility | 1.5 years
  Participants will report on perceptions of the study protocol in a post-intervention qualitative joint couple interview that utilizes a semi-structured couple interview guide. The guide includes specific prompts focused on recruitment, randomization, and assessments.
  In addition to these qualitative data collected from participants, data on recruitment feasibility will also be collected with an item on the contact form potential participants complete. Data on assessment feasibility will also be collected based on completion of measures and the length of time participants spend on these measures at each assessment.

SECONDARY OUTCOMES:
Physical activity. | 1.5 years
  Assessed pre/post-intervention with the International Physical Activity Questionnaire (IPAQ)-Long and a 7-day accelerometer assessment. Assessed monthly with the IPAQ-7 day. Participants will also self-report minutes of moderate-to-vigorous physical activity over the past week at each attended intervention class.
  IPAQ questionnaires assess self-reported walking, moderate intensity, and vigorous intensity physical activity as well as overall sedentary time. Accelerometers provide objective assessments of these constructs.
Diet. | 1.5 years
  Assessed pre/post-intervention with the Automated Self-Administered 24-hr diet assessment from the NCI (ASA-24). The ASA is a detailed 24-hour recall of food including portion sizes and preparation.
  Assessed pre/post-intervention and monthly during the intervention with the Rapid Eating Assessment for Participants- Shortened Version (REAP-S), a brief measure of diet quality and content over an average week.
Sleep. | 1.5 years
  Assessed pre/post-intervention and monthly with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance 8a item scale (SD) and the PROMIS Sleep-Related Impairment 8a item scale (SRI). Participants will also self-report their daily sleep during the 7-day pre/post-intervention accelerometer wear.
  The SD assesses sleep quality with 8 statements including "my sleep was restless," and the SRI assesses the impact of poor sleep and sleepiness on daily behaviors with 8 statements including "I had problems during the day because of poor sleep." Item responses on both measures range from 1 (not at all) to 5 (very much).
BMI | 1.5 years
  Weight in kilograms and height in meters will be measured pre-intervention by Clinical Research Unit staff in order to calculate BMI.
Waist circumference | 1.5 years
  Waist circumference in inches will be measured pre-intervention by Clinical Research Unit staff.
Weight | 1.5 years
  Weight in kilograms will be assessed pre-intervention by Clinical Research Unit staff and weight in pounds will also be collected before each intervention class by Lifestyle Coaches.
  Weight in pounds will be collected post-intervention with a medical-grade scale.
Blood glucose. | 1.5 years
  Assessed at pre-intervention by Clinical Research Unit medical staff: fasting blood glucose, HbA1c, 2-hr post glucose load (following 75 g OGTT).
  Assessed at post-intervention by the A1c Now point-of-care system test: HbA1c.
Anxiety. | 1.5 years
  Assessed pre/post-intervention and monthly with the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 8a item scale. This 8-item measure includes statements such as "I felt fearful."
Depression. | 1.5 years
  Assessed pre/post-intervention and monthly with the PROMIS Depression 8a item scale, which includes 8 statements such as "I felt worthless."
Affect. | 1.5 years
  Participants will complete the Positive and Negative Affective Scale (PANAS) daily during the pre/post-intervention 7-day accelerometer wear. The PANAS assesses positive and negative affect over the last day with 20 items. Participants rate from 1 (very slightly to none at all) to 7 (extremely) the extent to which they experienced each item (e.g., "nervous") in the past day.
Relationship satisfaction. | 1.5 years
  Assessed pre/post-intervention and monthly with the 16-item Couples Satisfaction Index (CSI), a measure of overall relationship satisfaction. Assessed daily during the pre/post-intervention 7-day accelerometer wear using a brief 4-item version of the CSI.
Partner support. | 1.5 years
  Assessed pre/post-intervention and at months 3, 6, 9 during the intervention, with the Social support and Exercise Survey and the Social Support and Eating Habits Survey. These measures assess the amount of support individuals seeking to exercise regularly perceive from family members and the amount of support individuals seeking to improve their diet receive from family members.
  Participants will also report on daily emotional and instrumental support during the pre/post-intervention 7-day accelerometer wear.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine JW Baucom, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguirre MC, Brown H, Gershenoff D, Hinton KL, Huntzinger OM, Klein N, Ramos C, Tavake-Pasi OF, Witte B, Wolfsfeld M, Sher T, Simmons DL, Smith TW, Clark L, Baucom KJW. The Role of Advocacy in Adapting the Diabetes Prevention Program for Couple-Based Delivery That Reaches Marginalized Groups. Behav Ther (N Y N Y). 2020 Oct;43(7):261-265. No abstract available. PMID 33536698
- [Background] Whitaker M, Aguirre MC, Gutierrez Chavez M, Beaulieu E, Arones YB, Gershenoff D, Hinton K, Klein N, Munezerou Uwizeye J, Napia E, Ramos C, Tavake-Pasi OF, Villalta J, Wolfsfeld C, Witte B, Maxfield E, Raphael K, Simmons DL, Clark L, Sher T, Smith TW, Baucom KJ. Couple-based lifestyle intervention to prevent type 2 diabetes: protocol for a randomised pilot trial. BMJ Open. 2023 Feb 16;13(2):e068623. doi: 10.1136/bmjopen-2022-068623. PMID 36797025

DOCUMENTS (1):
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT05695170/ICF_001.pdf